CLINICAL TRIAL: NCT01673633
Title: Sacroiliitis in Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Didem Arslan Tas, Internist and rheumatologist, Cukurova University
Other Study IDs: Sacroiliitis in SSc; 05/01/2012-4/21 (Other: 05/01/2012-4/21)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Systemic Sclerosis; Sacroiliitis; Inflammatory Back Pain
MeSH Terms: conditions — Scleroderma, Systemic; Sacroiliitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- SSc: Sacroiliitis
- Rheumatoid arthritis: Sacroiliitis
- Healthy controls: Sacroiliitis

SUMMARY:
One of the major problems of systemic sclerosis (SSc) patients is suggested to be articular involvement. Mostly involved joints in SSc were reported as wrist, carpometacarpal-interphalangeal, foot, knee, hip and shoulder however there have been little knowledge on sacroiliac joint. Here the investigators plan a study on the involvement of this joint in SSc.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as systemic sclerosis and rheumatoid arthritis and healthy volunteers

Exclusion Criteria:

* Not giving informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive systemic sclerosis and rheumatoid arthritis patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2012-01

PRIMARY OUTCOMES:
The frequency of sacroiliitis in systemic sclerosis | One year